CLINICAL TRIAL: NCT03826316
Title: A Study to Evaluate Pharmacokinetics of Nalbuphine Hydrochloride (10 mg/mL) After a Single Intravenous Administration in Healthy Volunteers Under Fasting Conditions
Brief Title: Pharmacokinetics of Nalbuphine Injection
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yung Shin Pharm. Ind. Co., Ltd. (Industry)
Collaborators: Taichung Veterans General Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: YSP-RJH3002-01
Record Dates: First submitted 2019-01-27; First posted 2019-02-01 (Actual); Last update posted 2019-02-01 (Actual); Status verified 2019-01

CONDITIONS: Pain, Postoperative
Keywords: Pharmacokinetic
MeSH Terms: conditions — Pain, Postoperative | interventions — Nalbuphine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mutonpain Injection 10 mg/ml (Experimental)
  Interventions: Drug: Nalbuphine

INTERVENTIONS:
Drug: Nalbuphine — Pharmacokinetic study under fasting conditions

SUMMARY:
A study to evaluate pharmacokinetics of nalbuphine hydrochloride (10 mg/mL) after a single intravenous administration in healthy volunteers under fasting conditions

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult male subjects between 20-45 years of age.
2. Body weight within 80-120% of ideal body weight.

   * Ideal body weight (kg) = [height (cm) - 80] *0.7 for male subjects
3. Acceptable medical history and physical examination including:

   * no particular clinically significant abnormalities in chest x-ray and electrocardiogram results within six months prior to study drug dosing.
   * no particular clinical significance in general disease history within two months prior to study drug dosing.
4. Acceptable biochemistry determinations (within normal limits or considered by the investigator or physician to be of no clinical significance) within two months prior to study drug dosing, which includes Serum Glutamic Oxaloacetic Transaminase (SGOT, same as AST), Serum Glutamic Pyruvic Transaminase (SGPT, same as ALT), Gamma-Glutamyl-Transpeptidase (γ-GT), alkaline phosphatase, total bilirubin, albumin, glucose, Blood Urea Nitrogen(BUN), uric acid, creatinine, total cholesterol and triglyceride (TG).
5. Acceptable hematology (within normal limits or considered by the investigator or physician to be of no clinical significance) within two months prior to study drug dosing, which includes hemoglobin, hematocrit, red blood cell count, white blood cell count with differentials and platelets.
6. Acceptable urinalysis (within normal limits or considered by the investigator or physician to be of no clinical significance) within two months prior to study drug dosing, which includes power of hydrogen (pH), blood, glucose, ketones, bilirubin and protein.
7. Male subjects willing to use a condom during any sexual contact with females of reproductive potential for up to 10 weeks after study drug dosing.
8. Have signed the written informed consent to participate in the study.

Exclusion Criteria:

1. A clinically significant disorder involving the cardiovascular, respiratory, hepatic, renal, gastrointestinal, immunologic, hematologic, endocrine or neurologic system(s) or psychiatric disease (as determined by the investigator).
2. A clinically significant illness or surgery within four weeks prior to dosing (as determined by the investigator).
3. History of gastrointestinal obstruction, inflammatory bowel disease, gallbladder disease, pancreas disorder over last two years or history of gastrointestinal tract surgery over last five years.
4. History of kidney disease or urination problem over last two years deemed by the investigator to be clinically significant.
5. Known or suspected history of drug abuse within lifetime as judged by the investigator.
6. History of alcohol addiction or abuse within last five years as judged by the investigator.
7. History of allergic response(s) to nalbuphine hydrochloride or any other related drugs.
8. Evidence of chronic or acute infectious disease.
9. Positive results for serum hepatitis B surface antigen (HBsAg), hepatitis C antibody (HCVAb), or human immunodeficiency virus (HIV).
10. Female subjects demonstrating a positive pregnancy screen prior to the study.
11. Female subjects who are currently breastfeeding.
12. Taking any drug known to induce or inhibit hepatic drug metabolism within four weeks prior to dosing. Examples of inducers include: piperidines, carbamazepine, dexamethasone and rifampin. Examples of inhibitors include: cimetidine, diphenhydramine, fluvastatin, methadone and ranitidine.
13. Taking any prescription medications within four weeks or any nonprescription medications (excluding flu vaccination) within two weeks prior to dosing.
14. Use of any investigational drug within four weeks prior to dosing.
15. Donating more than 250 milliliter (mL) of blood within two months prior to dosing or donating plasma (e.g. plasmapheresis) within two weeks prior to dosing.
16. Any other medical reason as determined by the investigator.

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2018-01-15 (Actual); Primary Completion 2018-11-22 (Actual); Study Completion 2019-01-15 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration (AUC) | Plasma sample: 0, 0.5, 5, 10, 15, 20, 30, 45 minutes, 1, 2, 4, 6, 8, 10 and 12 hours
Peak Drug Concentration (Cmax) | Plasma sample: 0, 0.5, 5, 10, 15, 20, 30, 45 minutes, 1, 2, 4, 6, 8, 10 and 12 hours
Elimiation half-life (T1/2) | Plasma sample: 0, 0.5, 5, 10, 15, 20, 30, 45 minutes, 1, 2, 4, 6, 8, 10 and 12 hours
Area under the (first) moment plasma concentration-time curve (AUMC) | Plasma sample: 0, 0.5, 5, 10, 15, 20, 30, 45 minutes, 1, 2, 4, 6, 8, 10 and 12 hours

SECONDARY OUTCOMES:
Adverse events | Adverse event reporting will up to 10 weeks.

CONTACTS AND LOCATIONS:
Locations (1):
- Taichung Veterans General Hospital, Taichung, Taiwan